CLINICAL TRIAL: NCT02467439
Title: Acute Partner and Social Contact Referral: iKnow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-2869; UNCPM 21414 (Other: UNC); 1R01AI114320-01 (NIH)
Record Dates: First submitted 2015-05-29; First posted 2015-06-10 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Acute HIV Infection; HIV Seropositive; Sexually Transmitted Infections
Keywords: unaware intervention;; contract sexual partner referral; peer referral
MeSH Terms: conditions — HIV Seropositivity; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Notification Cards (Active Comparator): Includes two groups of newly diagnosed HIV-infected participants (ppt): Seropositive and Acutely Infected. After consent and a full survey, blood and urine sample are collected for viral genetic testing and future STI testing. Ppts will be given notification cards for their sexual partners, social contacts. Ppts will receive contract partner notification: if the named sexual partners do not present for testing within 7-14 days, community outreach workers will contact and counsel the partners to visit the clinic. Any returning sexual partner or social contact presenting to the clinic with the notification card linking to the original index ppt will be consented (HIV testing, blood and urine specimen collected for viral genetic testing and future STI testing if HIV positive). If HIV-infected, they will be in the active arm, and will receive partner notification and social contact referral cards. If they are HIV-seronegative they will be screened for acute HIV infection.
  Interventions: Other: Notification cards
- Base Case Arm (No Intervention): consist of HIV seropositive and seronegative STI clinic patrons . After a brief survey to obtain demographics and sexual behavior, seronegative ppts will have blood collected for screening for acute HIV infection. If a person has acute HIV infection, they will be contacted by a community outreach worker and brought back in for counseling, and, if consenting, enrolled in the active arm. STI clinic patrons who are seropositive at screening will be given cards and asked to refer their sexual partners for evaluation using passive referral. Sexual partners presenting to the clinic with the notification card linking to the original index ppt in the base case arm will be consented to be in study (HIV testing, blood and urine specimen collected for viral genetic testing and future STI testing if HIV positive). If they are seropositive, these participants will be in the base case arm, and will receive partner notification cards for passive referral.

INTERVENTIONS:
Other: Notification cards — detection of AHI, contract partner notification, and social contact referral to find persons unaware of their HIV infection.
  Arms: Notification Cards

SUMMARY:
The primary purpose of this research is to assess the benefit of an "unaware intervention package" for identifying high risk persons who are unaware of their HIV infection status. This intervention package includes screening for acute HIV infection, contract sexual partner referral, and peer referral.

DETAILED DESCRIPTION:
This two-arm randomized study will evaluate an "unaware intervention package" among HIV-infected persons attending Sexually Transmitted Infection (STI) clinics in Lilongwe, Malawi. The package includes detection of Acute HIV Infection (AHI), contract partner notification, and social contact referral to find persons unaware of their HIV infection. The package will be compared to the current standard of care, passive partner notification, as the base case. Participants will be randomized to receive the intervention package - classified as the "active arm" of the study. The study will characterize the HIV stage (acute, recent, chronic) of the index participants and their sexual partners and social contacts, and use the HIV staging combined with sexual behavior data, phylogenetic analyses, and egocentric sexual/social network assessments to assess the potential impact of the intervention on ongoing transmission. We will obtain the distributions of numerous transmission-related attributes among the recruited contacts/partners of STI clinic patients, including contacts' and partners' HIV infection status and stage, HIV diagnosis/care/treatment status, STI status, and sexual behaviors. This information will allow us to model testing, linkage, and treatment interventions targeted to the traced partners and/or social contacts of acute, recent, and/or chronic index cases identified in STI clinics. We can then assess and compare the predicted effects on population-level HIV incidence of interventions attached to each recruitment method (tracing partners, social contacts, or both) and index case and contact disease stage (acute, recent, and/or chronic).

ELIGIBILITY:
Inclusion Criteria:

* Active and Base Case Index Participants:

  * Acute HIV-1 infection documented by a negative or discordant rapid HIV test results and detectable HIV RNA OR established HIV infection based on two positive HIV antibody rapid tests at the time of screening.
  * Men and women age >/= 18 years.
  * Current resident in the Lilongwe area.
  * Ability and willingness of participant to provide informed consent.
  * Willingness to provide contact/locator information to be contacted for AHI results if rapid test is negative or discordant.

Partners and Social Contacts (referred by active arm):

* Referred by active arm participant and presenting to STI clinics with a referral card.
* Men and women age >/= 18 years.
* Intention to remain in the Lilongwe area for the duration of the study.
* Ability and willingness of participant to provide informed consent.
* Willingness to provide contact/locator information to be contacted for AHI results if rapid test is negative or discordant.

Partners (referred by base case arm):

* Referred by base case arm participant and presenting to STI clinics with a referral card.
* Men and women age >/= 18 years.
* Ability and willingness of participant to provide informed consent.

Exclusion Criteria:

Active and Base Case Index Participants:

* HIV-negative based on one or more antibody rapid test and an HIV RNA PCR test.
* Serious illness, including tuberculosis or opportunistic infection, requiring systemic treatment and/or hospitalization.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Any other condition that in the opinion of the study investigator would compromise the safety of the study participant or study staff, or would prevent proper conduct of the study.

Partner and Social Contacts (referred by active or base case arm):

* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness, including tuberculosis or opportunistic infection, requiring systemic treatment and/or hospitalization.
* Any other condition that in the opinion of the study investigator would compromise the safety of the study participant or study staff, or would prevent proper conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15310 (Actual)
Dates: Start 2015-06; Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
the proportion of HIV-seropositive index participants with at least one newly diagnosed HIV-infected partner or social contact | 4 years

SECONDARY OUTCOMES:
The proportion of HIV-seropositive index participants with at least one HIV-infected person referred who is not in care (newly diagnosed plus known diagnoses not in care) | 4 years
Total HIV-infected persons, including all subsequent referrals, referred per first-wave index | 4 years
Total number of sexual partners referred (sexual partners or social contacts) per index | 4 years
Total number of persons referred per index. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: William Miller, MD, PhD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Kimberly Powers, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Maierhofer CN, Powers KA, Matoga MM, Chen JS, Jere E, Massa C, Mmodzi P, Bhushan NL, Phiri S, Hoffman IF, Lancaster KE, Miller WC, Rutstein SE. Characterizing Network-Based HIV Testing Interventions to Guide HIV Testing and Contact Tracing at STI Clinics in Lilongwe, Malawi. J Acquir Immune Defic Syndr. 2023 Oct 1;94(2):151-159. doi: 10.1097/QAI.0000000000003240. PMID 37345996
- [Derived] Chen JS, Matoga M, Pence BW, Powers KA, Maierhofer CN, Jere E, Massa C, Khan S, Rutstein SE, Phiri S, Hosseinipour MC, Cohen MS, Hoffman IF, Miller WC, Lancaster KE. A randomized controlled trial evaluating combination detection of HIV in Malawian sexually transmitted infections clinics. J Int AIDS Soc. 2021 Apr;24(4):e25701. doi: 10.1002/jia2.25701. PMID 33929094